CLINICAL TRIAL: NCT06936137
Title: : EFFECT OF PROBIOTIC SUPPLEMENTATION ON ATYPICAL ANTIPSYCHOTIC INDUCED WEIGHT GAIN IN PATIENTS ATTENDING PSYCHIATRIC CLINICS AT AINSHAMS UNIVERSITY HOSPITALS (A RANDOMIZED CONTROLLED TRIAL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD343/2024
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Antipsychotic Induced Weight Gain
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic supplementation (Lacteol fort 10 billion) which contains culture medium and lactobacillus (Experimental)
  Interventions: Drug: lactobacillus LS
- Participants will be advised to be adherent to their standard treatment and followed up regularly. (No Intervention)

INTERVENTIONS:
Drug: lactobacillus LS — Probiotic supplementation (Lacteol fort 10 billion) which contains culture medium and lactobacillus LS as active ingredients
  Arms: Probiotic supplementation (Lacteol fort 10 billion) which contains culture medium and lactobacillus

SUMMARY:
the goal of the study is to improve the quality of life of patients on antipsychotic medications and increase the rate of compliance to treatment.

Primary objective:

1.To determine the effectiveness of probiotics to decrease the weight gained as a result of antipsychotic medications.

Secondary objective:

1. To determine the effect of probiotic supplementation on the psychological state of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult schizophrenia patients (18-45 years) on second generation antipsychotics Stable patients with a total positive and negative syndrome scale (PANSS) score of ≤60.

With more than 10% weight gain after taking atypical antipsychotics for at least 3 months with treatment duration not more than two years.

Exclusion Criteria:

1. Taking probiotics, fiber supplements, antibiotics and laxatives in the last 6 weeks.
2. Comorbid gastrointestinal diseases, including active peptic ulcer, uncontrolled and recurrent diarrhea, gastrointestinal bleeding, and digestive system neoplastic diseases.

   -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of probiotics to decrease the weight gained as a result of antipsychotic medications. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university hospitals, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided